CLINICAL TRIAL: NCT04465331
Title: Adaptation and Validation of the Exercise Adherence Rating Scale of Knee Osteoarthritis Patients
Brief Title: Adaptation and Validation of the Exercise Adherence Rating Scale of Knee Osteoarthritis Patients (GONEARS)
Acronym: GONEARS
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2019 COUDEYRE 2; 2019-A01680-57 (Other: ANSM)
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Physical activity; Questionnaire; Adhesion
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity; Tissue Adhesions | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with knee arthrosis: Painful Knee Osteoarthritis with presence of osteophytes on radiography
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — completion of Exercise Adherence Rating Scale (EARS)

SUMMARY:
The origin of knee osteoarthritis is multifactorial but the disease is strongly related to age. The pain and functional disability are the main reasons for consultation. Non-pharmaceutical treatment is always indicated.

The rehabilitation will reduce the pain, maintain or partially recover the amplitude of the movements as well as fight against vicious analgesic attitudes and strengthen the muscles to stabilize the joints. A program of self-rehabilitation exercises performed at home may be prescribed to people with knee osteoarthritis. It must include exercises adapted to the patient's functional abilities and painful level and requires education to improve the patient's motivation to practice a regular exercise program. However, adherence to such exercises is low, and until 2016 there was no objective way to find out the reasons for patients' lack of adherence to self-workout programs. The EARS ("Exercise Adherence Rating Scale" or Adhesion to Physical Exercise Programs) is validated in 2016 and reliable to evaluate the physical activity of patients with low back pain.

As far as we know, this questionnaire is the only one validated in the international literature, a validation for French patients is currently underway. We believe this tool can be used for patients with knee osteoarthritis after minor changes.

DETAILED DESCRIPTION:
EARS ("Exercise Adherence Rating Scale" or Adhesion to Physical Exercise Programs) assesses in the first part what type of physical exercise was recommended for patients with common chronic pain, as well as their frequencies and the date until which they were prescribed. The patient can also inform how often he can do his exercises, or otherwise, if he has completely stopped them, to mention since when and why.

A second part of the questionnaire explores the behavior of patients towards adherence to exercise programs and a final part examines the reasons for or not performing these exercises.

Inclusion and the first questionnaires period at the beginning of the knee rehabilitation program (program for 6 weeks). Clinical and demographic data questionnaire that will be completed by the investigating physician. The second questionnaire will be done at 48 hours from the inclusion (only the EARS questionnaire will be filled at 2 days). The third time the patients will complete the questionnaires at the end of the rehabilitation program and the last time at 4 months end half.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Painful Knee Osteoarthritis with presence of osteophytes on radiography
* At least 1 of the following 3 criteria's: adult >50 years old, morning stiffness <30 minutes, or in the pre-stage surgical (programmed knee prosthesis replacement).
* Acceptance to participate in the study
* Patients affiliated to a social security scheme (beneficiary entitled)

Exclusion Criteria:

* Patient under guardianship, or protection of justice.
* Cognitive impairment
* Contraindications to Physical Activities
* Patient in the incapacity to answer the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Painful Knee Osteoarthritis with presence of osteophytes on radiography
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Assessment of adherence to physical exercise programs | Day 0
  measured by Exercise Adherence Rating Scale (EARS)
Assessment of adherence to physical exercise programs measured by Exercise Adherence Rating Scale (EARS) | Day 2
  measured by Exercise Adherence Rating Scale (EARS)
Assessment of adherence to physical exercise programs measured by Exercise Adherence Rating Scale (EARS) | Day 45
  measured by Exercise Adherence Rating Scale (EARS)
Assessment of adherence to physical exercise programs measured by Exercise Adherence Rating Scale (EARS) | Day 135
  measured by Exercise Adherence Rating Scale (EARS)

SECONDARY OUTCOMES:
knowledge of emotional state measured by questionnaire HAD (Hospital Anxiety and Depression Scale ) | Day 0
  The Hospital Anxiety and Depression Scale (HADS) is a valid and reliable self-rating scale that measures anxiety and depression in both hospital and community settings. HADS gives clinically meaningful results as a psychological screening tool and can assess the symptom severity and caseness of anxiety disorders and depression in patients with illness and the general population.
  One questionnaire, comprising fourteen questions. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
  Scoring : 0-7- normal, 8-10-borderling abnormal, 11-21-abnormal
knowledge of emotional state measured by questionnaire HAD (Hospital Anxiety and Depression Scale ) | Day 45
  The Hospital Anxiety and Depression Scale (HADS) is a valid and reliable self-rating scale that measures anxiety and depression in both hospital and community settings. HADS gives clinically meaningful results as a psychological screening tool and can assess the symptom severity and caseness of anxiety disorders and depression in patients with illness and the general population.
  One questionnaire, comprising fourteen questions. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
  Scoring : 0-7- normal, 8-10-borderling abnormal, 11-21-abnormal
knowledge of emotional state measured by questionnaire HAD (Hospital Anxiety and Depression Scale ) | Day 135
  The Hospital Anxiety and Depression Scale (HADS) is a valid and reliable self-rating scale that measures anxiety and depression in both hospital and community settings. HADS gives clinically meaningful results as a psychological screening tool and can assess the symptom severity and caseness of anxiety disorders and depression in patients with illness and the general population.
  One questionnaire, comprising fourteen questions. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
  Scoring : 0-7- normal, 8-10-borderling abnormal, 11-21-abnormal
personal efficacy by means of the questionnaire ASES "Arthritis Self-Efficacy Scale" | Day 0
  The ASES includes 20 questions that represent three subscales: pain, function, and other symptoms. Score ranging : from 1 to 10 (higher = greater self-efficacy).
personal efficacy by means of the questionnaire ASES "Arthritis Self-Efficacy Scale" | Day 45
  The ASES includes 20 questions that represent three subscales: pain, function, and other symptoms. Score ranging : from 1 to 10 (higher = greater self-efficacy).
personal efficacy by means of the questionnaire ASES "Arthritis Self-Efficacy Scale" | Day 135
  The ASES includes 20 questions that represent three subscales: pain, function, and other symptoms. Score ranging : from 1 to 10 (higher = greater self-efficacy).
Patient Global Impression of Change by Scale (PGIC) | Day 45
  This scale evaluates all aspects of patients' health and assesses if there has been an improvement or decline in clinical status. It consists of one item.
  Patient choose: 1 -No change (or condition has gotten worse), 2 - Almost the same, hardly any change at all, 3 - A little better, but no noticeable change, 4 - Somewhat better, but the change has not made any real difference, 5 - Moderately better, and a slight but noticeable change, 6 - Better and a definite improvement that has made a real and worthwhile difference, 7 - A great deal better and a considerable improvement that has made all the difference.
Patient Global Impression of Change by Scale (PGIC) | Day 135
  This scale evaluates all aspects of patients' health and assesses if there has been an improvement or decline in clinical status. It consists of one item.
  Patient choose: 1 -No change (or condition has gotten worse), 2 - Almost the same, hardly any change at all, 3 - A little better, but no noticeable change, 4 - Somewhat better, but the change has not made any real difference, 5 - Moderately better, and a slight but noticeable change, 6 - Better and a definite improvement that has made a real and worthwhile difference, 7 - A great deal better and a considerable improvement that has made all the difference.
Knee injury and Osteoarthritis Outcome Score (KOOS) | Day 45
  This scale evaluates all aspects the patients' opinion (symptoms, functional disability in activities of daily life or sports activities, quality of life) about their knee and hip problems, both for traumatic and degenerative joint diseases
Knee injury and Osteoarthritis Outcome Score (KOOS) | Day 135
  This scale evaluates all aspects the patients' opinion (symptoms, functional disability in activities of daily life or sports activities, quality of life) about their knee and hip problems, both for traumatic and degenerative joint diseases
The perceived barriers to and facilitators of physical activity | Day 45
  5. The perceived barriers to and facilitators of physical activity are measured by EPAP
The perceived barriers to and facilitators of physical activity | Day 135
  5. The perceived barriers to and facilitators of physical activity are measured by EPAP

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Coudeyre, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France